CLINICAL TRIAL: NCT02096614
Title: Multi-center, Investigator Initiated Phase 1 Study of MAGE-A4 Specific TCR Gene Transferred T Lymphocytes With Solid Tumors
Brief Title: Investigator Initiated Phase 1 Study of TBI-1201
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mie University (Other)
Collaborators: Takara Bio Inc. (Industry); Shionogi (Industry); Fiverings Co., Ltd. (Other); Statcom Co. Ltd. (Unknown)
Responsible Party: Principal Investigator, Shinichi Kageyama, Professor, Mie University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1201-01
Record Dates: First submitted 2014-03-19; First posted 2014-03-26 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Solid Tumors
Keywords: Adoptive cell transfer; Cell therapy; Immunotherapy; MAGE-A4; Esophageal cancer; Melanoma; Head and neck cancer; Ovarian cancer; TCR gene therapy
MeSH Terms: conditions — Esophageal Neoplasms; Melanoma; Head and Neck Neoplasms; Ovarian Neoplasms | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Low dose TBI-1201 with pre-treatment 1 (Experimental): TBI-1201(5*10^8) single-dose administration with pre-treatment of cyclophosphamide alone.
  Interventions: Drug: TBI-1201; Drug: Cyclophosphamide
- High dose TBI-1201 with pre-treatment 1 (Experimental): TBI-1201(5*10^9) single-dose administration with pre-treatment of cyclophosphamide alone.
  Interventions: Drug: TBI-1201; Drug: Cyclophosphamide
- High dose TBI-1201 with pre-treatment 2 (Experimental): TBI-1201(5*10^9) single-dose administration with pre-treatment of cyclophosphamide and fludarabine.
  Interventions: Drug: TBI-1201; Drug: Cyclophosphamide; Drug: Fludarabine
- TBI-1201 with pre-treatment 1 or 2 (Experimental): Arm1, 2 or 3, which is considered as optimal.
  Interventions: Drug: TBI-1201; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Drug: TBI-1201 — TBI-1201(5*10^8 or 5*10^9) is administered.
  Other Names: MAGE-A4-specific TCR gene transduced T lymphocytes
Drug: Cyclophosphamide — Cyclophosphamide (750mg/m2/day x 2 days Intravenous (IV)) is administered as pre-treatment medication of TBI-1201
  Other Names: Endoxan
Drug: Fludarabine — Fludarabine (20mg/m2 x 5 days Intravenous(IV)) is administered as pre-treatment medication of TBI-1201 in combination with cyclophosphamide.
  Other Names: Fludara
  Arms: High dose TBI-1201 with pre-treatment 2; TBI-1201 with pre-treatment 1 or 2

SUMMARY:
Following pre-treatment with cyclophosphamide and/or fludarabine, MAGE-A4-specific TCR gene transduced T lymphocytes are transferred to the patients with MAGE-A4-expressing solid tumors.

DETAILED DESCRIPTION:
Following pre-treatment with cyclophosphamide alone or in combination with fludarabine, MAGE-A4-specific TCR gene transduced T lymphocytes are transferred to HLA-A*24:02 positive patients with solid tumors which are 1) unresectable, refractory to standard therapy (chemotherapy, radiotherapy, etc), metastatic or recurrent, and 2) MAGE-A4-expressing. The primary objective is to evaluate the safety and in vivo kinetics, and the secondary is to evaluate clinical effect.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed solid tumors
2. Solid tumor, which is unresectable , refractory to standard therapy (chemotherapy, radiotherapy, etc) , metastatic or recurrent
3. HLA-A*24:02 positive
4. MAGE-A4-expression by PCR or immunohistochemistry
5. ECOG Performance Status, 0 or 1
6. Age >20 years on consent
7. No treatment (surgery, chemotherapy, radiotherapy, etc.) and expected sufficient recovery from the treatment at the time of the lymphocytes collection for gene transfer.
8. Life expectancy >= 16 weeks after consent
9. No severe damage on the major organs (bone marrow, heart, lung, liver, kidney, etc) and meet the following lab value criteria:

   * WBC > 2,500/μL
   * Hemoglobin > 8.0g/dL
   * Platelets > 75,000/μL
   * T. bilirubin < 1.5 x ULN
   * AST(GOT)、ALT(GPT) < 3.0 x ULN
   * Creatinine < 1.5 x ULN
10. Ability to understand the study contents and to give a written consent at his/her free will.

Exclusion Criteria:

1. The following serious complications are excluded from the study;

   * Unstable angina, cardiac infarction, or heart failure
   * Uncontrolled diabetes or hypertension
   * Active infection
   * Obvious interstitial pneumonia or lung fibrosis by chest X-ray
   * Active autoimmune disease requiring steroids or immunosuppressive therapy
2. Serious hypersensitivity
3. Tumor cell invasion into CNS
4. Active multiple cancer
5. Positive for HBs antigen/antibody, HBc antibody, or HCV antibody, and virus DNA observed in serum, except for HBs antibody positive case who had vaccine injection before.
6. Positive for antibodies against HIV or HTLV-1
7. Left Ventricular Ejection Fraction (LVEF): =< 50％
8. Percutaneous Oxygen saturation: < 94％
9. History of hypersensitivity reactions to bovine or murine derived substances.
10. History of hypersensitivity reaction to drugs used in this study
11. Psychological disorder or drug dependency which may have impact on the consent.
12. Pregnant females, lactating females (except when they cease and don't resume lactation) or female and male patients who cannot agree to practice the adequate birth control after the consent during the study
13. Clinically significant systemic illness that in the judgment of the PI or sub-investigator would compromise the patient's ability to tolerate protocol therapy or significantly increase the risk of complications.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-04; Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Incidence and grade of adverse events (CTCAE) | 8 weeks
  Confirm the toxicity profile, which is measured by the degree of grade and seriousness, duration, causality, classification, etc. of the adverse events.
Appearance of replication competent retrovirus by PCR | 8 weeks
  Confirm no replication competent retrovirus observed
Appearance of clonality by LAM-PCR | 8 weeks
  Confirm no clonality is observed
Kinetics of TBI-1201 in blood by realtime-PCR and flow cytometry | 8 weeks
  Evaluate persistence and expansion of transferred TBI-1201

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Shiku, M.D., Ph.D., Study Chair — Department of Immuno-Gene Therapy, Mie University, graduate School of Medicine; Shinichi Kageyama, M.D., Ph.D., Principal Investigator — Mie University Hospital
Locations (1):
- Mie University Hospital, Tsu, Mie-ken, Japan